CLINICAL TRIAL: NCT02354300
Title: A Prospective Study of the Treatment of Intracranial Aneurysms Using Pipeline Flow-Diverter Embolization in Conjunction With Transcranial Dopplers (TCD)
Brief Title: Transcranial Doppler Ultrasound Monitoring During Flow-Diverter Embolization
Status: Completed | Type: Observational
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Other Study IDs: 201400923
Record Dates: First submitted 2015-01-29; First posted 2015-02-03 (Estimated); Last update posted 2016-08-26 (Estimated); Status verified 2016-08

CONDITIONS: Intracranial Aneurysm; Aneurysm, Intracranial; Giant Intracranial Aneurysm
MeSH Terms: conditions — Intracranial Aneurysm

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- TCD Ultrasound: Transcranial doppler ultrasound monitoring during flow diverter placement.
  Interventions: Device: TCD Ultrasound

INTERVENTIONS:
Device: TCD Ultrasound — Transcranial doppler ultrasound monitoring will occur during flow diverter placement.
  Other Names: TCD

SUMMARY:
Flow diverters have been approved since 2012 for the treatment of large, wide neck intracranial aneurysms. These devices have been associated with embolic events which cause blockage in a blood vessel and can result in long term complications. One possible cause of these events is the formation of small emboli during placement of the device.

DETAILED DESCRIPTION:
Flow diverters have been developed to treat intracranial aneurysms. Embolisms have occurred in a small percentage of patients which can result in long term complications including stroke, hemorrhage, and even death.

The formation of microemboli during the insertion of the device has not been evaluated. During insertion, there is significant disruption of blood flow and this may be a source of intracranial microemboli.

This study will use transcranial doppler ultrasound (TCD) to evaluate the blood flow during the placement of flow diverters to try to determine why these embolic events occur.

ELIGIBILITY:
Inclusion Criteria:

* Adult subjects 18 years of age and older
* Non-pregnant
* Diagnosis of intracranial aneurysm that will be clinically treated with a flow diverter

Exclusion Criteria:

* Pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Outpatient clinic
Sampling Method: Non-Probability Sample
Enrollment: 2 (Actual)
Dates: Start 2015-04; Primary Completion 2015-04 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Occurence of microemboli | 1 day
  The number of subjects who experience microemboli during device placement.

CONTACTS AND LOCATIONS:
Overall Officials: Spiros Blackburn, MD, Principal Investigator — University of Florida
Locations (1):
- University of Florida, Gainesville, Florida, United States

IPD SHARING:
Plan to Share IPD: No